CLINICAL TRIAL: NCT00039338
Title: Randomized Phase III Study Of Neoadjuvant Chemotherapy Followed By Surgery Vs. Concomitant Radiotherapy And Chemotherapy In FIGO Ib2, IIa>4 cm or IIb Cervical Cancer
Brief Title: Chemotherapy Followed By Surgery Vs Radiotherapy Plus Chemotherapy in Patients With Stage IB or II Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55994; 2008-003396-52 (EudraCT Number)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer; stage IIB cervical cancer; stage IIA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy; Brachytherapy; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy followed by surgery (Experimental): neoadjuvant chemotherapy (Cisplatin) followed by surgery (radial hysterectomy)
  Interventions: Procedure: conventional surgery; Procedure: neoadjuvant chemotherapy; Drug: cisplatin
- Radio-chemotherapy (Active Comparator): Concomitant radiotherapy (external radiotherapy combined with external boost or brachytherapy) and chemotherapy (cisplatin)
  Interventions: Procedure: neoadjuvant chemotherapy; Radiation: brachytherapy; Radiation: radiation therapy; Drug: cisplatin

INTERVENTIONS:
Procedure: conventional surgery — Radial hysterectomy
  Arms: Chemotherapy followed by surgery
Procedure: neoadjuvant chemotherapy — Experimental arm: minimal cumulative cisplatin dose of 225 mg/m2. Comparator arm: cumulative cisplatin dose of 200-240 mg/m2.
Radiation: brachytherapy — Brachytherapy at the end of external radiation. Minimal total dose (external with or without external boost + brachytherapy) of 75 Gy EQD2 to point A. Overall treatment less than 50 days.
  Arms: Radio-chemotherapy
Radiation: radiation therapy — Between 45-50 Gy, in fractions of 1.8 to 2 Gy.
  Arms: Radio-chemotherapy
Drug: cisplatin — Minimal cumulative 225 mg/m2 (experimental arm). Cumulative 200-240 mg/m2 (comparator arm).

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed during surgery. Radiation therapy uses high-energy x-rays to kill tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known whether chemotherapy is more effective followed by surgery or combined with radiation therapy in treating cervical cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy followed by radical hysterectomy with that of chemotherapy plus radiation therapy in treating patients who have stage IB or stage II cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall and progression-free survival of patients with stage IB2, IIA, or IIB cervical cancer treated with neoadjuvant cisplatin-based chemotherapy followed by radical hysterectomy vs standard therapy comprising concurrent radiotherapy and cisplatin-based chemotherapy.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, FIGO stage, age (18 to 50 vs 51 to 75), and histological subtype (adenomatous vs non-adenomatous component). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive neoadjuvant cisplatin-based chemotherapy on day 1. Treatment repeats every 21 days. Within 6 weeks after the last chemotherapy course, patients undergo a type III-V Piver-Rutledge radical hysterectomy. Patients with positive lymph nodes or tumor invasion into the parametria or less than 5 mm from the resection borders after surgery receive standard adjuvant external beam radiotherapy once daily, 5 days a week, for 5-5.6 weeks (25-28 treatment days) followed by external boost radiotherapy or brachytherapy for 1 or 2 days.
* Arm II: Patients receive standard therapy comprising radiotherapy as in arm I concurrently with cisplatin-based chemotherapy once weekly for 6 weeks. Adjuvant hysterectomy is allowed, but not recommended, in case of histologically proven residual tumor.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity. For patients in both arms, cisplatin may be combined with other chemotherapeutics as long as the minimum platinum dose is given.

Quality of life is assessed at baseline and at 6, 12, 18, and 24 months.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 686 patients (343 per treatment arm) will be accrued for this study within 3.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical cancer, including the following subtypes:

  * Squamous cell carcinoma
  * Adenosquamous cell carcinoma
  * Adenocarcinoma (excluding small cell, clear cell, and other rare variants of the classical adenocarcinoma)
* FIGO stage IB2, IIA (greater than 4 cm), or IIB

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.46 mg/dL

Renal:

* Creatinine clearance greater than 60 mL/min

Other:

* No other prior or concurrent malignancy except adequately treated basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent anticancer agent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2002-03; Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Landoni, MD, Study Chair — Istituto Europeo Di Oncologia, Milano; Alessandro Colombo, MD, Study Chair — Ospedale Alessandro Manzoni, Lecco; Stefano Greggi, MD, PhD, Study Chair — Istituto Nazionale per lo Studio e la Cura dei Tumori, Napoli; Gemma G. Kenter, MD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam
Locations (24):
- Austria (2):
  - Karl-Franzens-University Graz, Graz
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
- Centre Regional Francois Baclesse, Caen, France
- Italy (6):
  - Istituto Europeo Di Oncologia, Milan
  - Ospedale San Gerardo, Monza
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori, Naples
  - Ospedale Mauriziano Umberto I, Torino
  - Clinica Universitaria, Turin
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (7):
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Erasmus MC - Daniel den Hoed Cancer Center, Rotterdam
  - Universitair Medisch Centrum - Academisch Ziekenhuis, Utrecht
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Hospital Universitario San Carlos, Madrid, Spain
- United Kingdom (3):
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Mid Kent Oncology Centre, Maidstone, Kent

REFERENCES:
- [Derived] Kenter GG, Greggi S, Vergote I, Katsaros D, Kobierski J, van Doorn H, Landoni F, van der Velden J, Reed N, Coens C, van Luijk I, Colombo N, Steen-Banasik EV, Ottevanger N, Casado A; EORTC-55994 Study Group. Randomized Phase III Study Comparing Neoadjuvant Chemotherapy Followed by Surgery Versus Chemoradiation in Stage IB2-IIB Cervical Cancer: EORTC-55994. J Clin Oncol. 2023 Nov 10;41(32):5035-5043. doi: 10.1200/JCO.22.02852. Epub 2023 Sep 1. PMID 37656948